CLINICAL TRIAL: NCT04172259
Title: A Multi-center Randomized Phase II Study of Doxorubicin Liposome Versus Epirubicin Plus Cyclophosphamide Combined With Trastuzumab and Pertuzumab(HP), Followed by Taxon Plus HP as Neoadjuvant Therapy for HER2-positive Early Breast Cancer
Brief Title: ACHP-THP vs EC-THP as Neoadjuvant Therapy for HER2-positive EBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xia Wen, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METIS; SCBCG-023 (Other: South China Breast Cancer Group)
Record Dates: First submitted 2018-12-18; First posted 2019-11-21 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy
Keywords: Human epidermal growth factor receptor 2; Pathology complete response
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; 1-dodecylpyridoxal; Cyclophosphamide; Trastuzumab; Docetaxel; Epirubicin; pertuzumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACHP-THP (Experimental): Doxorubicin liposome（PLD）35 mg/m2 Cyclophosphamide（CTX）600 mg/m2 Trastuzumab：first cycle 8mg/kg，then 6mg/kg Pertuzumab：first cycle 840mg，then 420mg Docetaxel（DOC）75 mg/m2 every 3 weeks paclitaxel (PTX) 175 mg/m2 every 3 weeks or paclitaxel (PTX) 80 mg/m2 every week albumin-bound paclitaxel 260 mg/m2 or albumin-bound paclitaxel 100 mg/m2 every week
  Interventions: Drug: Doxorubicin liposome; Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Docetaxel; Drug: Pertuzumab; Drug: Paclitaxel-albumin
- EC-THP (Active Comparator): Epirubicin（EPI）90 mg/m2 Cyclophosphamide（CTX）600 mg/m2 Trastuzumab：first cycle 8mg/kg，then 6mg/kg Pertuzumab：first cycle 840mg，then 420mg Docetaxel（DOC）75 mg/m2 every 3 weeks paclitaxel (PTX) 175 mg/m2 every 3 weeks or paclitaxel (PTX) 80 mg/m2 every week albumin-bound paclitaxel 260 mg/m2 or albumin-bound paclitaxel 100 mg/m2 every week
  Interventions: Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Docetaxel; Drug: Epirubicin; Drug: Pertuzumab; Drug: Paclitaxel; Drug: Paclitaxel-albumin

INTERVENTIONS:
Drug: Doxorubicin liposome — PLD
  Other Names: PLD
  Arms: ACHP-THP
Drug: Cyclophosphamide — CTX
  Other Names: CTX
Drug: Trastuzumab — H
  Other Names: Herceptin
Drug: Docetaxel — DOC
  Other Names: Taxotere
Drug: Epirubicin — EPI
  Other Names: EPI
  Arms: EC-THP
Drug: Pertuzumab — P
Drug: Paclitaxel — paclitaxel (PTX) 175 mg/m2 every 3 weeks or paclitaxel (PTX) 80 mg/m2 every week
  Arms: EC-THP
Drug: Paclitaxel-albumin — albumin-bound paclitaxel 260 mg/m2 or albumin-bound paclitaxel 100 mg/m2 every week

SUMMARY:
Breast cancer is the most common malignant tumor in women. EC-TH is one of the standard chemotherapy regimens for HER-2 positive early breast cancer(EBC). Earlier use of trastuzumab may improve DFS rate. In this study, the investigators want to find out whether ACH-TH regimen compared with the EC-TH regimen in HER2+ EBC could improve the pCR rate in neoadjuvant chemotherapy.

We update protocol in Sep 2020, because Pertuzumab is approveled by Chinese goverment and coverd by national insurance, dual target therapy with Trastuzumab and Pertuzumab is the standard therapy for neoadjuvant therapy of HER2-positive EBC patients.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women. EC-TH is one of the standard chemotherapy regimens for HER-2 positive early breast cancer(EBC). Earlier use of trastuzumab could improve the DFS rate in HER2+ EBC. But due to the cardio-toxicity of both anthracycline and trastuzumab, the investigators usually avoid using these two drugs synchronously. The guidelines do not recommend ECH-TH regemin because of cardiac adverse effect. Doxorubicin liposome(A) has equivalent effect as anthracycline in advaced breast cancer(ABC), lower cardiac toxicity and could be combined use with trastuzumab. In this study, the investigators want to find out whether ACH-TH regimen compared with the EC-TH regimen in HER2+ EBC could improve the pCR rate in neoadjuvant chemotherapy.

We update protocol in Sep 2020, because Pertuzumab is approveled by Chinese goverment and coverd by national insurance, dual target therapy with Trastuzumab and Pertuzumab is the standard therapy for neoadjuvant therapy of HER2-positive EBC patients. So now we want to compare ACHP-THP regimen compared with the EC-THP regimen in HER2+ EBC could improve the pCR rate in neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age, </= 70 years of age.
* HER2-positive breast cancer
* Histologically confirmed invasive breast carcinoma
* Clinical stage T2-4/N0-3/M0 or node positive at presentation (patients with T1 tumors will not be eligible)
* Known hormone-receptor status
* Non previous anti-breast cancer neoadjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic, renal and liver function
* Screening Left ventricular ejection fraction (LVEF) >/= 50% on echocardiogram (ECHO)
* Adequate organ function

Exclusion Criteria:

* Stage IV (metastatic) breast cancer or bilateral breast cancer
* History of any prior (ipsi- or contralateral breast cancer except lobular carcinoma in situ)
* History of other malignancy within the last 5 years except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other non-breast malignancies with a similar outcome to those mentioned above
* Cardiopulmonary dysfunction as defined by protocol
* Current severe, uncontrolled systemic disease
* Pregnant or lactating women
* Any known active liver disease, e.g. due to HBV, HCV, autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent serious uncontrolled infections requiring treatment or known infection with HIV
* History of intolerance, including Grade 3 to 4 infusion reaction or
* hypersensitivity to trastuzumab or chemotherapy drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response rate (pCR) | At the time of definitive surgery (approximately 24-36 weeks from first dose of study drug).
  Pathological complete response (pCR) in the breast tissue and the lymph node tissue will be assessed upon completion of pre-operative systemic therapy and definitive surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 20-24 weeks from first dose of study drug
  CRR is defined as the proportion of subjects with complete or partial radiographic response of the primary tumor as determined by the central imaging vendor.
Event Free Survival (EFS) | Up to 5 years from the date of definitive surgery
  EFS will be defined as the time from random assignment to documentation of the first of the following events: discontinuation of study therapy due to protocol-defined progression prior to surgery; local, regional, or distant recurrence of breast cancer following curative surgery; a new breast cancer; another new onset malignancy; or death as a result of any cause.
Overall Survival (OS) | Up to 5 years from the date of definitive surgery.
  OS will be defined as the number of days from the day the subject is randomized to the date of the subject's death.
Incidence of chemotherapy-induced cardiotoxicity | Approximately 20-24 weeks from first dose of study drug
  Incidence of chemotherapy-induced cardiotoxicity, according to NCI-CTCAE 4.03 version.
Change From Baseline Between Treatment Comparison in Euro Quality of Life (EQ-5D) Index | First day of treatment (Day 1) up to 6 months during the post-surgery follow-up period (approximately 15 months from first dose of study drug)
  The EuroQol EQ-5D is a 6-item instrument designed to assess health status in terms of a single index value or utility score. It contains 5 descriptors of current health state (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 3 levels of function (1=no problem, 2=some problem, and 3=extreme problem). The scores on the 5 descriptors are summarized to create a single summary score. An overall utility score is calculated based on these domains, with a range score from 0 (worse health scenario) to a maximum of 1.0 (best health scenario).
Change From Baseline Between Treatment Comparison in Functional Assessment of Cancer Therapy -Breast (FACT-B) | First day of treatment (Day 1) up to 6 months during the post-surgery follow-up period (approximately 15 months from first dose of study drug)
  FACT is a modular approach to assess participant health-related quality of life using a 'core' set of questions (FACT-G) as well as a cancer site-specific module. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The FACT-B consisted of the FACT-G (27-item) and a breast-specific module: a 10-item instrument designed to assess participant concerns relating to breast cancer. For all questions, participants were asked to respond to a five-level scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. FACT-B total score = Physical Well-Being + Social/Family Well-Being + Emotional Well-Being + Functional Well-Being + Breast Cancer Subscale. As each of the items ranges from 0-4, the range of possible scores is 0-144, with 0 being the worst possible score and 144 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xia, MD, Principal Investigator — SunYat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Fisher B, Gunduz N, Saffer EA. Influence of the interval between primary tumor removal and chemotherapy on kinetics and growth of metastases. Cancer Res. 1983 Apr;43(4):1488-92. PMID 6831397
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Goldie JH, Coldman AJ. A mathematic model for relating the drug sensitivity of tumors to their spontaneous mutation rate. Cancer Treat Rep. 1979 Nov-Dec;63(11-12):1727-33. PMID 526911
- [Background] Adjuvant Pertuzumab and Trastuzumab in Early HER2-Positive Breast Cancer. N Engl J Med. 2017 Aug 17;377(7):702. doi: 10.1056/NEJMx170011. Epub 2017 Jul 12. No abstract available. PMID 28700263
- [Background] Martin M, Holmes FA, Ejlertsen B, Delaloge S, Moy B, Iwata H, von Minckwitz G, Chia SKL, Mansi J, Barrios CH, Gnant M, Tomasevic Z, Denduluri N, Separovic R, Gokmen E, Bashford A, Ruiz Borrego M, Kim SB, Jakobsen EH, Ciceniene A, Inoue K, Overkamp F, Heijns JB, Armstrong AC, Link JS, Joy AA, Bryce R, Wong A, Moran S, Yao B, Xu F, Auerbach A, Buyse M, Chan A; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in HER2-positive breast cancer (ExteNET): 5-year analysis of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1688-1700. doi: 10.1016/S1470-2045(17)30717-9. Epub 2017 Nov 13. PMID 29146401
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Background] Dieras V, Miles D, Verma S, Pegram M, Welslau M, Baselga J, Krop IE, Blackwell K, Hoersch S, Xu J, Green M, Gianni L. Trastuzumab emtansine versus capecitabine plus lapatinib in patients with previously treated HER2-positive advanced breast cancer (EMILIA): a descriptive analysis of final overall survival results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):732-742. doi: 10.1016/S1470-2045(17)30312-1. Epub 2017 May 16. PMID 28526536
- [Background] Krop IE, Kim SB, Martin AG, LoRusso PM, Ferrero JM, Badovinac-Crnjevic T, Hoersch S, Smitt M, Wildiers H. Trastuzumab emtansine versus treatment of physician's choice in patients with previously treated HER2-positive metastatic breast cancer (TH3RESA): final overall survival results from a randomised open-label phase 3 trial. Lancet Oncol. 2017 Jun;18(6):743-754. doi: 10.1016/S1470-2045(17)30313-3. Epub 2017 May 16. PMID 28526538
- [Background] Schneeweiss A, Chia S, Hickish T, Harvey V, Eniu A, Hegg R, Tausch C, Seo JH, Tsai YF, Ratnayake J, McNally V, Ross G, Cortes J. Pertuzumab plus trastuzumab in combination with standard neoadjuvant anthracycline-containing and anthracycline-free chemotherapy regimens in patients with HER2-positive early breast cancer: a randomized phase II cardiac safety study (TRYPHAENA). Ann Oncol. 2013 Sep;24(9):2278-84. doi: 10.1093/annonc/mdt182. Epub 2013 May 22. PMID 23704196
- [Background] Extra JM, Antoine EC, Vincent-Salomon A, Delozier T, Kerbrat P, Bethune-Volters A, Guastalla JP, Spielmann M, Mauriac L, Misset JL, Serin D, Campone M, Hebert C, Remblier C, Bergougnoux L, Campana F, Namer M. Efficacy of trastuzumab in routine clinical practice and after progression for metastatic breast cancer patients: the observational Hermine study. Oncologist. 2010;15(8):799-809. doi: 10.1634/theoncologist.2009-0029. Epub 2010 Jul 29. PMID 20671105
- [Background] Perez EA, Suman VJ, Davidson NE, Gralow JR, Kaufman PA, Visscher DW, Chen B, Ingle JN, Dakhil SR, Zujewski J, Moreno-Aspitia A, Pisansky TM, Jenkins RB. Sequential versus concurrent trastuzumab in adjuvant chemotherapy for breast cancer. J Clin Oncol. 2011 Dec 1;29(34):4491-7. doi: 10.1200/JCO.2011.36.7045. Epub 2011 Oct 31. PMID 22042958
- [Background] Jankowitz RC, Brufsky AM. Adjuvant treatment of HER2-positive breast cancer: winning efforts continue to improve HER2-positive patient outcome long-term. Breast Cancer Res. 2012 Apr 30;14(2):308. doi: 10.1186/bcr3120. PMID 22546039
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846
- [Background] Rafiyath SM, Rasul M, Lee B, Wei G, Lamba G, Liu D. Comparison of safety and toxicity of liposomal doxorubicin vs. conventional anthracyclines: a meta-analysis. Exp Hematol Oncol. 2012 Apr 23;1(1):10. doi: 10.1186/2162-3619-1-10. PMID 23210520
- [Background] Wolff AC, Wang M, Li H, Pins MR, Pretorius FJ, Rowland KM, Sparano JA, Davidson NE. Phase II trial of pegylated liposomal doxorubicin plus docetaxel with and without trastuzumab in metastatic breast cancer: Eastern Cooperative Oncology Group trial E3198. Breast Cancer Res Treat. 2010 May;121(1):111-20. doi: 10.1007/s10549-010-0838-7. Epub 2010 Mar 24. PMID 20333545
- [Background] Martin M, Sanchez-Rovira P, Munoz M, Baena-Canada JM, Mel JR, Margeli M, Ramos M, Martinez E, Garcia-Saenz JA, Casado A, Jaen AM, Gonzalez-Farre X, Escudero MJ, Rodriguez-Martin C, Carrasco E; GEICAM. Pegylated liposomal doxorubicin in combination with cyclophosphamide and trastuzumab in HER2-positive metastatic breast cancer patients: efficacy and cardiac safety from the GEICAM/2004-05 study. Ann Oncol. 2011 Dec;22(12):2591-2596. doi: 10.1093/annonc/mdr024. Epub 2011 Mar 17. PMID 21421542
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986